CLINICAL TRIAL: NCT07171034
Title: A Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of KLA318-2 Nanocrystal Injection in Healthy Participants
Brief Title: A Phase I Study of KLA318-2 Nanocrystal Injection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hunan Kelun Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KLA318-2-101
Record Dates: First submitted 2025-08-28; First posted 2025-09-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: Healthy
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- KLA318-2 Nanocrystal Injection 60mg (Experimental): 12 participants receive KLA318-2 60mg
  Interventions: Drug: KLA318-2 Nanocrystal Injection
- KLA318-2 Nanocrystal Injection 120mg (Active Comparator): Period 1, 6 participants receive KLA318-2 120mg → 6 participants receive Celebrex Capsule 200mg; Period 2, 6 participants receive Celebrex Capsule 200mg → 6 participants receive KLA318-2 120mg
  Interventions: Drug: KLA318-2 Nanocrystal Injection; Drug: Celebrex Capsule
- KLA318-2 Nanocrystal Injection 180mg (Active Comparator): Period 1, 6 participants receive KLA318-2 180mg → 6 participants receive Celebrex Capsules 400mg; Period 2, 6 participants receive Celebrex Capsules 400mg → 6 participants receive KLA318-2 180mg
  Interventions: Drug: KLA318-2 Nanocrystal Injection; Drug: Celebrex Capsule
- KLA318-2 Nanocrystal Injection 240mg (Experimental): 12 participants receive KLA318-2 240mg
  Interventions: Drug: KLA318-2 Nanocrystal Injection

INTERVENTIONS:
Drug: KLA318-2 Nanocrystal Injection — Intravenous injection, single dose
Drug: Celebrex Capsule — P.O., single dose
  Arms: KLA318-2 Nanocrystal Injection 120mg; KLA318-2 Nanocrystal Injection 180mg

SUMMARY:
The purpose of this study is to evaluate the safety,tolerability and pharmacokinetics properties of KLA318-2 Nanocrystal Injection after a single intravenous injection in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Health participants (Age: 18~45 years);
2. Body Weight: Male≥50.0kg, Female≥45.0kg; 18.5 ≤BMI≤ 28.0;
3. Normal ECG, showing no clinically relevant deviations, as judged by the investigator.

Exclusion Criteria:

1. Allergy or Drug hypersensitivity;
2. Clinically significant Medical History;
3. Gastrointestinal ulcers or gastrointestinal bleeding;
4. History of any surgery within 4 weeks;
5. History of any Medication within 14 days;
6. History of any drug interactions with celecoxib within 30 days;
7. History of any clinical study within 3 months;
8. History of any vaccine within 1 month;
9. History of any drug abuse, or positive drugs of abuse test result;
10. Subjects with difficult venous blood collection/intolerance to venipuncture, or with a history of needle phobia/blood phobia;
11. Massive blood loss (> 200 mL) in the past 3 months;
12. Special requirements for diet;
13. Heavy smoker ( more than 3 cigarettes/day) within 3 months;
14. History of alcohol abuse,or heavy alcohol intake (more than 14 units a week) within 6 months, or positive alcohol test;
15. Heavy caffeine intake;
16. History of grapefruit, xanthine-rich foods intake within 7 days;
17. Female participants are pregnant or lactating;
18. History of unprotected sex within 2 weeks.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | UP to Day 14

SECONDARY OUTCOMES:
PK parameter Cmax | UP to Day 3
  Maximum peak plasma concentration (Cmax) after single dose and in a steady state after multiple doses
PK parameter Tmax | UP to Day 3
  Time of Cmax (Tmax) after single dose and in a steady state after multiple doses
PK parameter AUC0-t | UP to Day 3
  Area under the concentration-time curve (AUC0-t) from time zero to time "t" after single dose and in a steady state after multiple doses
PK parameter AUC0-∞ | UP to Day 3
  AUC from time zero to infinity (AUC0-∞) after single dose and in a steady state after multiple doses
PK parameter t1/2 | UP to Day 3
  Terminal-phase elimination half-life (t1/2) after single dose and in a steady state after multiple doses

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No